CLINICAL TRIAL: NCT04596501
Title: Susceptibility to Thrombosis in Post-menopausal Women- Influence of Exercise Training
Brief Title: Exercise Training and Thrombotic Risk in Post-menopausal Women
Acronym: TIME
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Copenhagen (Other)
Collaborators: Swansea University (Other)
Responsible Party: Principal Investigator, Ylva Hellsten, Professor, University of Copenhagen
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: Thrombosis in PM Women
Record Dates: First submitted 2020-10-08; First posted 2020-10-22 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Thrombosis; Menopause; Exercise Training; Vascular Dilation
MeSH Terms: conditions — Thrombosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early postmenopausal women (Experimental): Healthy sedentary early postmenopausal women
  Interventions: Other: Early and late postmenopausal women
- Late postmenopausal women (Experimental): Healthy sedentary late postmenopausal women
  Interventions: Other: Early and late postmenopausal women

INTERVENTIONS:
Other: Early and late postmenopausal women — The intervention involves supervised team sports 1 h 3 x/week for 16 weeks.

SUMMARY:
At menopausal transition, the risk of cardiovascular diseases increases. This is partly due to aging, but largely also the loss of estrogen, which has many positive effects on the circulation and protects against cardiovascular diseases. It has been suggested that the loss of estrogen may have a negative impact on the otherwise well-documented health promoting effects of exercise training, and that the time after menopause may be crucial for the effect of exercise training on the vascular function, and therefore also for the risk of thrombosis. Literature regarding the effect of exercise training on the risk of thrombosis is limited, and especially in women.

The purpose of the present study is to investigate whether the same effects of exercise training in relation to thrombosis is achieved if the exercise is initiated early compared to late after menopause. The aim is to provide knowledge-based recommendations regarding exercise. Teams sports will be used as the training intervention, because team sports benefits physical health and also includes a social element.

DETAILED DESCRIPTION:
Part of the novelty of this project is to link functional measurements of cardiovascular health at whole body level to cell studies. Cells will be isolated from muscle samples obtained from the post-menopausal women before and after the training intervention. This will enhance the understanding of the changes that occur after prolonged loss of estrogen on thrombotic risk and vascular function, and whether exercise training can alter these parameters.

ELIGIBILITY:
Inclusion Criteria:

* Age: 50-70 years
* Physical activity ≤ 2 hours per week (except transportation by bike or by walking)
* BMI ≤ 30

Exclusion Criteria:

* Age <50 years
* Injuries that prevent the performance of team sports
* Participation in other clinical projects
* Smokes or has smoked within the last 10 years
* On hormone therapy
* Not entered menopause
* Has chronic diseases that are not expected, cf. the groups sought. Including heart problems, atrial fibrillation, cancer, immune diseases and previous strokes with functionally significant sequelae
* Being treated with oral steroids
* Has alcohol / drug abuse or is being treated with disulfiram (Antabus)
* Is unable to understand the contents of the document with informed consent or the experimental procedures

Ages: 50 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in clot microstructure in early and late postmenopausal women after 16 weeks of exercise training | 16 weeks
  Clot microstructure is measured in a rheometer using unaltered whole blood
Changes in platelet reactivity in early and late postmenopausal women after 16 weeks of exercise training | 16 weeks
  Platelet reactivity is measured with Light Transmission Aggregometry using platelet rich and platelet poor plasma
Plasma concentration of coagulation factors in early and late postmenopausal women after 16 weeks of exercise training | 16 weeks
  Coagulation factors II, VII, X, VIII, D-dimer, fibrinogen and thrombin
Changes in vascular function in early and late postmenopausal women after 16 weeks of exercise training | 16 weeks
  Vascular function is assessed by flow-mediated dilation (FMD) in the brachial artery using ultrasound doppler
Changes in capillary density after 16 weeks of team sports in early and late postmenopausal women | 16 weeks
  Capillary density will be assessed by histochemistry
Changes in proliferative capacity of endothelial cells after 16 weeks of exercise training in early and late postmenopausal women | 16 weeks
  From a biopsy sample we isolate endothelial cells and run a proliferation assay
Changes in mitochondrial function of endothelial cells after 16 weeks of exercise training in early and late postmenopausal women | 16 weeks
  High resolution respirometry
Changes in skeletal muscle protein content important for vascular function after 16 weeks of exercise training in early and late postmenopausal women | 16 weeks
  Western blots will be used to determine endothelial nitric oxide synthase (eNOS), cyclo-oxygenase 1 and 2, prostacyclin synthase, endothelin receptor A and B, VEGF (vascular endothelial growth factor), Thrombospondin-1, Flk-1 (VEGF receptor). All protein content measures will be presented as arbitrary units.

SECONDARY OUTCOMES:
Changes in blood pressure after 16 weeks of team sports in early and late postmenopausal women | 16 weeks
  Blood pressure measured at home with an automated blood pressure device. Systolic blood pressure, diastolic blood pressure and mean arterial pressure will be collected.
Changes in maximal oxygen uptake after 16 weeks of team sports in early and late postmenopausal women | 16 weeks
  Maximal oxygen uptake will be measured using a metabolic cart. The test protocol will be performed on a cycle ergometer using an incremental step test.
Changes in body composition after 16 weeks of team sports in early and late postmenopausal women | 16 Weeks
  Dual-energy x-ray absorptiometry (DXA) will be used to determine fat free mass, fat mass as well as bone mineral content. These values will be presented in absolute (g) as well as relative values (percentage)

CONTACTS AND LOCATIONS:
Overall Officials: Ylva Hellsten, Dr.Med.Sci., Principal Investigator — Nutrition, Exercise and Sports, 2200 Copenhagen, Denmark
Locations (1):
- Ylva Hellsten, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No